CLINICAL TRIAL: NCT02590172
Title: Evaluation of the Methods and Effectiveness of Care for Eligible Medical and Surgical Patients on Admission in Continuous Monitoring Units
Acronym: UNISURC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI14008
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Units Continuous Monitoring (USC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In France, Intensive Medicine is carried out in three types of structures: intensive care units, intensive care unit and units Continuous Monitoring (USC). Created in the 90s as intermediate structures between conventional care units and intensive care units, these units are assigned to the care of patients whose conditions and treatment are fear the occurrence of one or more critical failures requiring to be monitored, or whose condition, at the end of one or more critical failure is too severe or unstable to allow a return to a classical inpatient unit.

Thus, USC represent a milestone in the journey of patients whose condition is critical: patients from the emergency services, patients in the immediate postoperative period, coming out of intensive care patients, or finally in conventional hospitalization patients whose condition s 'worse. The creation of the USC is not subject to authorization but must be contractualized between the hospital and the Regional Health Agency (ARS) because it is resource intensive. Organizations and their operating modes are guided by the recommendations of the French Society of Anesthesia and Intensive Care (SFAR), and the Society of French Language Resuscitation (SRLF) published in 2005.The US establishment has a beneficial effect on the quality of care and the care pathway of patients at risk shown by the reduction in morbidity and mortality, the rate of admission and / or USC readmission of length of stay and hospital stay costs.

It is possible to objectify provided first establish an inventory on the activity of these units and the patient base supported. To judge the benefit of the assumption by the USC, it is necessary to assess the adequacy of patients managed with an updated specification and defined by a group of experts.

DETAILED DESCRIPTION:
4600 adult patients will be enrolled in the study with the primary objective to quantify in terms of mortality reduction, "the benefit" of using USC on the effectiveness of the treatment and patient care pathway that present Medical eligibility criteria to supervision USC.

The methodology of the study is organized into 5 phases:

* Development of candidate criteria that justify the presence in USC and validation by a panel of experts according to the Delphi method
* Selection of a representative sample of 100 institutions with USC stratified by major regions (North, Ile-de-France, Southeast, Southwest), the activity of the USC (number admissions / year), method of financing the establishment, presence or absence of an operating theater.
* Observational Cohort study, prospective, multicenter. In each selected center will be collected the data during consecutive patients 1-2 weeks depending on the activity centers on USC sectors, post-operative, post-resuscitation and post emergency. Data collection will be done on the ground and from Medicalization Programme of Information Systems extraction . An external quality control will be organized on 10% of stays.
* Determination of eligibility for hospitalization USC will be conducted by a group of professionals representing different companies analysis in pairs and independently stays.
* Modelling and economic evaluation: development and validation of the score (ASIC Activity Score for Intermediate Care) and medico-economic analysis.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age> = 18 years) hospitalized in a facility selected during the investigation period:

or in one of the three evaluated healthcare pathways: 1 / out patient surgery postoperative period; 2 / downstream of hospital emergencies; 3 / downstream resuscitation (excluding return home and external transfer), it is recognized or not USC.

USC is present during the investigation period. Patient who read the Circular.

Exclusion Criteria:

* opposition to the data collection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be one of the selected schools and hospitals among those with a USC.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
hospital Mortality | seven days
  Quantify in terms of mortality reduction, "the benefit" of using USC on the effectiveness of the treatment and patient care pathway with existing medical eligibility criteria to supervision USC

SECONDARY OUTCOMES:
Score ASIC | seven days
  Develop a score justifying the eligibility of patients USC: ASIC score for Intermediate Care Activity Score
typology of admitted patients | seven days
  Describe the organization and activity of USC in France by representative sampling.
hospital stay duration | seven days
numbers of serious adverse events | seven days
Readmission and death rates | seven days

CONTACTS AND LOCATIONS:
Overall Officials: Beaussier Marc, PHD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôptal Saint Antoine, Paris, France

REFERENCES:
- [Derived] Misset B, Aegerter P, Boulkedid R, Alberti C, Baillard C, Guidet B, Beaussier M. Construction of reference criteria to admit patients to intermediate care units in France: a Delphi survey of intensivists, anaesthesiologists and emergency medicine practitioners (first part of the UNISURC project). BMJ Open. 2023 Jul 24;13(7):e072836. doi: 10.1136/bmjopen-2023-072836. PMID 37487677